CLINICAL TRIAL: NCT04720391
Title: Bone Metastases in neurOendocrine NEoplasms: naTural History, Prognostic Impact and Therapeutic Approach (MONET)
Acronym: MONET
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1436
Record Dates: First submitted 2021-01-20; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Bone Metastases; Neuroendocrine Neoplasm
Keywords: NET; NEC; Neuroendocrine tumors; Neuroendocrine carcinomas; Bisphosphonates
MeSH Terms: conditions — Neuroendocrine Tumors; Carcinoma, Neuroendocrine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective/prospective observational multicentric trial on patients with bone metastases from NENs.

General objectives:

* To trace on a national scale the frequency of bone metastases in patients with neuroendocrine neoplasm (NEN) and their clinical management.
* To correlate clinical and biological factors to clinical outcomes.
* To centralise and to make homogeneous clinical, pathological, instrumental and therapeutic information.
* To set up a database and to acquire biological material for studying predictive and prognostic biomarkers.

DETAILED DESCRIPTION:
Background, rationale and objectives:

On March 25th 2015 the Ethical Committee from IEO approved the academic study entitled "Bone metastases in neuroendocrine tumors (NETs): a survey on natural history, prognostic value and treatment approach", version 1.0 30-Jan-2015. This was a retrospective study led to report how the issue bone metastases from NETs was handle in real practice. Preliminary data related to 321 patients from 18 Italian centers were presented as a poster at the ESMO 2017 congress (Fazio et al. 448P) and they will be included in a manuscript to submit for publication in a peer-review journal. The current protocol regards the continuation of the retrospective analysis, starting since 2014, since the previous study required data collection up to 2013, and at the same time a multicenter prospective observational analysis on the topic.

Duration of the study The study will regard patients fulfilling the eligibility criteria from 2014 to 2021. Data analysis will be completed by the year 2021.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of NEN
* Instrumental and/or histological diagnosis of bone metastasis
* At least one year of follow-up from the diagnosis of bone metastasis

Exclusion Criteria:

* Small cell lung carcinoma
* MiNEN
* Non neuroendocrine neoplasm

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with bone metastases from NENs histologically proved.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 01/2021 - 12/2021
  Overall survival (OS) will be calculated from the date of BM diagnosis to the date of death
Influence of skeletal related events (SRE) on survival | 01/2021 - 12/2021
  Influence of skeletal related events (SRE) on overall survival (OS)
Correlation between SRE and time from bone metastasis and SRE, site of one metastases, number of bone metastases, morphology of bone metastases, LDH | 01/2021 - 12/2021
  To evaluate the correlation between SRE and time from bone metastasis and SRE, site of one metastases, number of bone metastases, morphology of bone metastases, LDH
Influence of the use of bisphosphonates or RANK-ligands | 01/2021 - 12/2021
  To evaluate the influence of the use of bisphosphonates or RANK-ligands on overall survival

SECONDARY OUTCOMES:
Correlation from bone metastases and age, gender, primary site, Ki-67, grade of differentiation | 01/2021 - 12/2021
  To evaluate the correlation between bone metastases and patients and tumor's features
Natural history (time between diagnosis of NEN and first diagnosis of bone metastasis, frequency and time to SRE, sites of bone metastases) | 01/2021 - 12/2021
  To describe the natural history time between diagnosis of NEN and first diagnosis of bone metastasis, frequency and time to SRE, sites of bone metastases
Radiological diagnosis (CT, MRI) | 01/2021 - 12/2021
  To describe the morphological features of bone metastases in patients with NEN
Functional diagnosis (68GaPET/CT-DOTA-peptide, 18FDGPET/CT) | 01/2021 - 12/2021
  To To describe the functional features of bone metastases in patients with NEN
Impact of antitumor therapy on bone metastases behavior | 01/2021 - 12/2021
  To describe the global impact of antitumor therapies on bone metastases behavior
Impact of supportive care | 01/2021 - 12/2021
  To describe the global impact of supportive care on overal survival

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Fazio, M.D., Ph.D., Study Chair — European Institute of Oncology, IEO, IRCCS; Francesca Spada, M.D., Ph.D., Principal Investigator — European Institute of Oncology, IEO, IRCCS
Locations (1):
- European Institute of Oncology, IEO, IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harding JJ, Abu-Zeinah G, Chou JF, Owen DH, Ly M, Lowery MA, Capanu M, Do R, Kemeny NE, O'Reilly EM, Saltz LB, Abou-Alfa GK. Frequency, Morbidity, and Mortality of Bone Metastases in Advanced Hepatocellular Carcinoma. J Natl Compr Canc Netw. 2018 Jan;16(1):50-58. doi: 10.6004/jnccn.2017.7024. PMID 29295881
- [Result] Grisanti S, Bianchi S, Locati LD, Triggiani L, Vecchio S, Bonetta A, Bergamini C, Conte P, Airoldi M, Merlano M, Carlini P, Ibrahim T, Rossetto C, Alfieri S, Pronzato P, Tonoli S, Maroldi R, Nicolai P, Resteghini C, Magrini SM, Berruti A. Bone metastases from head and neck malignancies: Prognostic factors and skeletal-related events. PLoS One. 2019 Mar 20;14(3):e0213934. doi: 10.1371/journal.pone.0213934. eCollection 2019. PMID 30893350